CLINICAL TRIAL: NCT03730220
Title: Induction of Labour in Norway: a Pilot for a Prospective National Audit
Brief Title: The Norwegian Induction Project: a Pilot for a Prospective National Audit
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); Førde Central Hospital (Other); Sykehuset Innlandet HF (Other); Helse Fonna (Other); Helse Nord (Industry); Haukeland University Hospital (Other); Helse Nord-Trøndelag HF (Other); Nordlandssykehuset HF (Other); Sorlandet Hospital HF (Other Government); Sykehuset Telemark (Other Government); Sykehuset i Vestfold HF (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Sykehuset Ostfold (Other); Helse Møre og Romsdal HF (Other Government); Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ingvil Krarup Sørbye, Consultant, Oslo University Hospital
Other Study IDs: 2018/1087
Record Dates: First submitted 2018-08-21; First posted 2018-11-05 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Induced; Birth; Delivery Complication; Indications for Care in Pregnancy; Labor; and Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Induction of labour

SUMMARY:
The worldwide rate of induction of labour has been steadily increasing over the last 15 years, a trend that is reflected in Norway.

The overall aim of this study is to identify disparities between delivery departments in Norway in regards to:

1. The overall rate of labour induction
2. Main indication for the induction of labour.
3. Induction methods used and protocols followed
4. Maternal and fetal outcomes in induced births

Methods:

Observational study. Registration of induction indication, methods and outcomes in induced women. Data will be collected prospectively during a period of 4 months from 21 Norwegian delivery units using a web-based standardized case record form.

DETAILED DESCRIPTION:
In 2000 the Norwegian national induction rate was 8.8% of all births, but this increased to 21.8% in 2016. The regional induction rate varies between counties, varying from 17.7% of all births in Nordland to 24.0% in Rogaland. Individual units could have an even wider variation. There are reports of a high rate of induction in primiparous women. In some units, local audits have noted that in 2016, over 27% of primiparous women had their labour induced. Labour inductions in primiparous women (Robson group 2a) may be associated with an increased likelihood of caesarean sections and operative vaginal delivery. An increased caesarean rate in primiparous women will have implications for subsequent pregnancies. In Hammerfest Hospital, the caesarean section rate in Robson group 2a was 37% in 2016.

In Norway, induction of labour is offered in approximately 50 obstetric units. There are national guidelines available for the induction of labour from the Norwegian Gynaecological Society and from the Department of Health. , These guidelines are not categorical and leave the decision for the specific method, or regimen for labour induction, up to the attending gynaecologist or local departments. Thus, the national protocols between departments vary considerably and women living in different regions of Norway do not have the same options for induction of labour.

The Norwegian situation reflects the international situation where multiple induction protocols exist. There is no consensus regarding the medical criteria for the identification of women for induction of labour, nor the induction methods or protocols used.

Aim

The overall aim of this study is to identify disparities between delivery departments in Norway in regards to:

1. The overall rate of labour induction
2. Main indication for the induction of labour.
3. Induction methods used and protocols followed
4. Maternal and fetal outcomes in induced births

Methods:

Observational study where we perform a prospective registration of induction indication, methods and outcomes in induced women on a common internet platform electronic case record form (e-CRF) through Service For Sensitive Data/Tjeneste For Sensitive Data (TSD), University of Oslo (UiO).

Participating centres

1. AHUS
2. Arendal
3. Bærum
4. Drammen
5. Førde
6. Gjøvik
7. Haugesund
8. Hammerfest
9. Haukeland
10. Levanger
11. Lillehammer
12. Nordland Sentralsykehus
13. OUS Ullevål
14. OUS Rikshospitalet
15. Sykehuset i Vestfold
16. Sykehuset i Telemark
17. Tromsø
18. Trondheim
19. Kristiansand
20. Stavanger
21. Sykehuset Østfold, Kalnes
22. Ålesund

Data registration and project management :

Establishing an e-CRF at Service For Sensitive Data/Tjeneste For Sensitive Data (TSD) University of Oslo (UiO) (which each participating centre can access online to register variables. Project leader will apply for ethics permission from the Regional Ethics Committee. Each participating centre will apply for database permission from the local Protector of Patient Records (Personvernansvarlig).

Ethical considerations:

The individual health staff responsible for patient care will provide information about the study in Norwegian and English following the medical decision (that is taken independent of this study) to induce the patient. The patient has the right to refuse participation in the study.

Project committee:

Ingvil Krarup Sørbye, Kevin Sunde Oppegaard, Anne Flem Jacobsen

International advisor: Professor Andrew D. Weeks, Department of Women's and Children's Health, Liverpool Women's Hospital, University of Liverpool, Crown Street, Liverpool, L8 7SS, UK.

ELIGIBILITY:
Inclusion Criteria:

* Induced women with no previous vaginal delivery
* Gestational age from 23+0 weeks
* Viable pregnancy at time of inclusion

Exclusion Criteria:

* Previous vaginal delivery

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Delivery units in Norway with a yearly number of births of >1000, or delivery units with <1000 births per year, but with a selected birthing population
Sampling Method: Non-Probability Sample
Enrollment: 1846 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Caesarean rate | Throughout the study period of 3 months
  Caesarean rate in induced women

SECONDARY OUTCOMES:
Time from induction to delivery | From start of medication/balloon until time of birth of baby
  Time from induction initiation to delivery of baby in minutes
Composite infant outcome | From time of delivery until time of discharge of patient from maternity unit
  Low Apgar score and/or transfer to NICU and/or low pH in umbilical artery
Uterine tachysystole during labour | From start of labour as defined by opening of partograph until time of birth of baby
  More than 5 contractions each 10 minutes and fetal tracing abnormality
Indication for induction of labour | Throughout the study period of 3 months
  Proportions of main indications for labour induction
Induction method used | Throughout the study period of 3 months
  Proportions of different induction methods/protocols used

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Oppegaard, PhD, MD, Study Director — Helse Nord, Hammerfest Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be available for sharing. Only aggregated data in the results will be made available. The Study Protocol, Statistical Analysis Plan, Patient Information Form and results will be made available. The results will be made available immediately following publication, with anyone who wishes to access the data. Proposals may be submitted up to 31.12.2025 following article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 31.12.2020-31.12.2025
Access Criteria: Personal application